CLINICAL TRIAL: NCT01613508
Title: A Randomized Clinical Trial of Direct Anterior Approach and Mini-Posterior Approach Total Hip Arthroplasty
Brief Title: A Randomized Study of Approaches in Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael J. Taunton, M.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-001341
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Total Hip Replacement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Direct Anterior Approach (Active Comparator): An oblique incision is made over the anterior margin of the tensor muscle. The fascia of the tensor muscle is identified and incised. The muscle is swept digitally laterally and a retractor is placed over the superior aspect of the femoral neck. The hip capsule is then incised and retracted.
  Interventions: Procedure: Direct Anterior Approach
- Mini-Posterior Approach (Active Comparator): The surgical approach involved a 7 to 9.5 cm incision along the posterior aspect of the femur starting at the tip of the greater trochanter and proceeding distally. The fascia of the gluteus maximus was split, and blunt dissection revealed the underlying abductor and external rotator musculature. The external rotators an the hip capsule were incised and preserved as one layer, with an attempt being made to preserve the insertion of the quadratus femoris on the femur. The hip was dislocated posteriorly and the femoral neck was cut in accordance with the preoperative plan.
  Interventions: Procedure: Mini-Posterior Approach

INTERVENTIONS:
Procedure: Direct Anterior Approach
  Arms: Direct Anterior Approach
Procedure: Mini-Posterior Approach
  Arms: Mini-Posterior Approach

SUMMARY:
The primary aim of the study is to compare the results of an established, successful procedure, which is total hip arthroplasty through a mini-posterior approach to a less studied - increasingly popular procedure, which is total hip replacement through the direct anterior approach utilizing the orthopedic table.

ELIGIBILITY:
Inclusion Criteria

1. Male or Female patients between 20 and 100 with unilateral osteoarthritis (DJD) who are surgical candidates for total hip arthroplasty
2. Study participants must be able to give informed consent.

Exclusion Criteria

1. Significant proximal femoral deformity (post SCFE, Perthes, DDH), acetabular dysplasia (ANY CROWE), inflammatory arthritis, septic arthritis, osteomyelitis, prior infection of hip joint, significant leg length discrepancy (> 4cm), osteoporosis, arthrodesis of the affected hip.
2. The presence of infections, highly communicable diseases, e.g. AIDS, active tuberculosis, venereal disease, hepatitis.
3. Significant neurological or musculoskeletal disorders or disease that may adversely affect normal gait or weight bearing.
4. Presence of previous prosthetic hip replacement device (any type).
5. Active Metastatic disease
6. Active major Psychiatric illness
7. Active Drug or alcohol abuse
8. BMI > 40.
9. Patients that are known to be pregnant
10. Actively failing contralateral hip replacement.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2013-01; Primary Completion 2017-12-31 (Actual); Study Completion 2018-02-27 (Actual)

PRIMARY OUTCOMES:
Activity monitors will be worn | Baseline to 1 year
  3 monitoring sensors will be worn by the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Taunton, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States